CLINICAL TRIAL: NCT06359522
Title: A Comparative Study of Medical Management vs Transcatheter PDA Occlusion Using Near-Infrared Spectroscopy
Brief Title: PDA Occlusion Using NIRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Norton Healthcare (Other)
Responsible Party: Principal Investigator, Scott Duncan, Professor, University of Louisville
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22.0334
Record Dates: First submitted 2024-03-11; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Organ Perfusion Determined by Using NIRS Post Transcatheter PDA Occlusion or Medical Closure of PDA

STUDY DESIGN:
Intervention Model Description: Patients who are being treated for PDA closure either via transcatheter occlusion or medical closure as part of routine care are eligible for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Trancatheter occlusion (Other): Patients who are being treated with transcatheter occlusion for PDA closure are eligible to participate in this study for NIRS monitoring.
  Interventions: Device: NIRS monitor
- Medical closure (Other): Patients who are being treated with tylenol or indomethacin for medical closure of their PDA are eligible to participate in this study for NIRS monitoring.
  Interventions: Device: NIRS monitor

INTERVENTIONS:
Device: NIRS monitor — NIRS monitoring data will be collected to determine organ perfusion.

SUMMARY:
Our study will be a prospective observational study of all patients in the Norton Children's Hospital NICU (Neonatal Intensive Care Unit) who undergo a transcatheter PDA occlusion or medical closure of PDA to compare the two populations regarding changes in organ perfusion determined by using NIRS monitoring to follow the regional saturation of oxygen (rSO2) of the cerebral and renal regions. We suspect that medical treatment will have no significant change in rSO2 as described in previous literature. We also suspect that transcatheter occlusion will have minimal effects on rSO2 and be comparable to medical therapy.

DETAILED DESCRIPTION:
Informed Consent will be obtained prior to initiation of the study protocol. NIRS Monitoring (Cerebral and Renal) will be placed with skin probes on the scalp and abdomen up to 24 hours prior to initiation of treatment either through medical therapy (Tylenol or indomethacin) or transcatheter occlusion. These values will be used to create an average baseline for the patient. NIRS will be left on during treatment/procedure and for 5 days after treatment to monitor any changes during or after treatment of the PDA. Changes will be compared to baseline readings.

NIRS monitoring will be done with INOVS 7100 Regional Oximeter from Medtronic (https://www.medtronic.com/covidien/en-us/products/cerebral-somatic-oximetry/invos-7100 system.html). Data collection will be done through chart review and pulling logged data from the NIRS monitoring unit. Data to be collected will include type of treatment, gestational age, patient birth weight, patient weight at time of treatment, and rSO2 (Cerebral and Regional) rSO2 variation will be addressed by calculating Coefficients of Variance at 5min epochs which has been shown to decrease the effects of normal variation.

Standardized time points will be compared between the two groups as follows:

* Data to be collected will include type of treatment, gestational age, patient birth weight, patient weight at time of treatment, and rSO2 (Cerebral and Regional)
* rSO2 variation will b e addressed by calculating Coefficients of Variance at 5min epochs which has been shown to decrease the effects of normal variation (10).
* Standardized time points will be compared between the two groups as follows:

  1. Baseline Levels: 24 hours prior to treatment
  2. During the Procedure: during initiation of procedure, 5min after device placed,10 min post device placement, 30min post device placement and 1 hour post placement
  3. Levels at 12 hours post treatment, until 48 hours post and then daily until monitoring is discontinued.
  4. Arterial O2 Saturations, FiO2 %, mode of ventilation will be recorded at the above time points as well and fractionated
* Statistician will analyze data collected

ELIGIBILITY:
Inclusion Criteria:

* Infants in the Norton Children's NICU with hsPDA deemed to require closure either through medical therapy or transcatheter occlusion by the primary NICU care team.
* Parents or Legal Guardian provide written consent for the infant to participate in this study

Exclusion Criteria:

* Infants with other hemodynamically significant congenital heart disease that could affect systemic blood flow

Ages: 0 Months to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Measure changes in rScO2 and SrO2 after TCPC of a PDA and compare to baseline readings. | Baseline through 48 hours post procedure and daily for 5 days
  NIRS cerebral and regional monitoring
Measure changes in rScO2 and SrO2 after medical closure of PDA with Tylenol. | Baseline through 48 hours post procedure and daily for 5 days
  NIRS cerebral and regional monitoring

SECONDARY OUTCOMES:
Compare rates of co-morbid conditions between the two groups such as but not limited to necrotizing enterocolitis, feedings intolerance, or failed to extubate within 5 days post treatment. | Baseline through 5 days post-treatment
  Medical outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Norton Children's Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided